CLINICAL TRIAL: NCT00814892
Title: A Phase II Trial to Determine the Safety, Tolerability and Efficacy of an Allogeneic Whole Cell Vaccine Administered With Autologous Myeloid Dendritic Cells to Patients With Non-Metastatic Androgen Independent Prostate Carcinoma
Brief Title: Vaccine Therapy in Treating Patients With Non-Metastatic Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to funding issues.
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC0554; MC0554 (Other: Mayo Clinic Cancer Center); 06-004659 (Other: Mayo Clinic - IRB)
Record Dates: First submitted 2008-12-24; First posted 2008-12-25 (Estimated); Results first posted 2013-08-29 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-10

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DC-APCC (Experimental): Patients undergo standard leukapheresis to harvest peripheral blood mononuclear cells for dendritic cell vaccine preparation. Patients receive the APCC vaccine and autologous dendritic cells derived from CD14-positive myeloid peripheral blood cells ID on days 0, 14, and 28 and then every 28 days for up to 14 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: allogeneic tumor cell vaccine; Biological: therapeutic autologous dendritic cells

INTERVENTIONS:
Biological: allogeneic tumor cell vaccine — Given intradermally
Biological: therapeutic autologous dendritic cells — Given intradermally

SUMMARY:
RATIONALE: Vaccines made from tumor cells or dendritic cells may help the body build an effective immune response to kill tumor cells. It is not yet known which vaccine is more effective in treating patients with prostate cancer.

PURPOSE: This phase II trial is studying how well the combination of a proven effective allogenic whole prostate carcinoma cell (APCC) vaccine co-administered with ex vivo generated dendritic cells (DCs)(DC-APCC) extend the time to prostate cancer progression.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the proportion of patients with androgen-independent prostate cancer who are progression-free at one year after treatment with DC-APCC.

Secondary

* Evaluate treatment toxicity.
* Evaluate time to prostate-cancer specific mortality.
* Evaluate progression-free survival.
* Evaluate time to PSA progression, and duration of PSA-based response.
* Evaluate quality of life of patients treated with this regimen.

OUTLINE: Patients undergo standard leukapheresis to harvest peripheral blood mononuclear cells for dendritic cell vaccine preparation and will receive the APCC vaccine and autologous dendritic cells derived from CD14-positive myeloid peripheral blood cells ID in every 2 weeks for the first 2 treatments (cycle 1 and 2), and then every 4 weeks therafter for up to 14 administrations in the absence of disease progression or unacceptable toxicity. The first four patients will be observed for four weeks following the third DC-APCC vaccination to assess toxicity, the enrollment of patients will continue if toxicity related events not present.

Patients undergo blood sample collection periodically for translational studies. Samples are measured for a number of immune parameters by quantifying T-cell and dentritic cell populations by analysis of surface marker molecules by flow cytometry, T-cell proliferation assay, non-specific cytokine release, lysate-specific cytokine release, and cytokine expression measured by cytometric bead array and qPCR.

Patients complete quality-of-life questionnaires periodically.

After completion of study treatment, patients are followed periodically for up to 3 years.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Biochemically progressive disease defined by two serial PSA measurements obtained ≥ 1 week apart during ongoing optimal androgen-deprivation therapy (e.g., orchiectomy, luteinizing hormone-releasing hormone [LHRH] agonist, or another equivalent hormonal agent)

    * Concurrent LHRH agonist or high-dose bicalutamide required (unless patient has undergone prior orchiectomy)
* Has undergone prior standard primary therapy for prostate cancer (e.g., radical prostatectomy, radiotherapy, or an equivalent initial treatment directed towards localized prostate cancer)
* PSA 2.0-100.0 ng/mL
* Serum testosterone < 50 ng/dL (unless undergoing antiandrogen monotherapy)
* No concurrent evidence of radiological or new clinically palpable metastatic cancer

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 12 weeks
* WBC ≥ 3,500/µL
* Platelet count ≥ 100,000/µL
* Hemoglobin ≥ 10.0 g/dL
* Creatinine ≤ 2.0 mg/dL
* Alkaline phosphatase ≤ 2.5 times upper limit of normal (ULN)
* AST ≤ 2.5 times ULN
* Fertile patients must use effective contraception
* Willing to provide blood samples for research purposes
* Able to complete questionnaire(s) alone or with assistance
* Able to undergo leukapheresis
* No known immunodeficiency
* No other malignancy within the past 5 years except basal cell or squamous cell carcinoma of the skin treated with local resection only
* No concurrent serious illness
* No known history of positive PPD skin test

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* More than 1 month since prior and no concurrent corticosteroids or other immunosuppressive agents

  * Inhaled corticosteroids allowed
* More than 1 month since prior and no concurrent estrogens and/or ketoconazole
* More than 3 months since prior and no other concurrent investigational medicinal products
* More than 4 weeks since prior and no concurrent secondary hormonal maneuver with or without a peripheral antiandrogen (e.g., bicalutamide), PC-SPES, or any other herbal medicines used to treat prostate cancer
* No prior prostate cancer vaccine
* No other therapy for prostate cancer (e.g., chemotherapy, immunotherapy, radiotherapy, or new hormonal therapy) during and for 4 months after completion of study therapy
* No other concurrent standard therapy that is potentially curative or proven capable of extending life expectancy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish Kohli, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic Cancer Center, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two (2) participants were recruited between Jan 2009 and March 2010 at Mayo Clinic. This trial was permanently closed in March 2010 due to funding issues. Since only two participants were accrued, patient confidentiality prevents the reporting of these two participants.
Period: Overall Study
Arm/Group | DC-APCC
Started | 2
Completed | 0
Not Completed | 2
Not completed — Disease Progression | 1
Not completed — Study Termination | 1

BASELINE CHARACTERISTICS:
Population: Since only two participants were accrued, patient confidentiality prevents the reporting of these two participants.
Arm/Group | DC-APCC
Number analyzed (Participants) | 0
Age, Categorical [Count of Participants; unit: Participants]
Age Continuous [Mean (Standard Deviation); unit: years]
Sex: Female, Male [Count of Participants; unit: Participants]
Region of Enrollment [Number; unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Are Progression Free at One Year
Description: Progression free was defined as being free of radiographically detectable disease/metastases at one year after registration and having a prostate-specific antigen (PSA) level <200.0 ng/mL.
Time Frame: One year
Population: Since only two participants were accrued, patient confidentiality prevents the reporting of these two participants.
Arm/Group | DC-APCC
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Severe Adverse Events
Description: Severe adverse events were defined as grade 3 or higher, regardless of attribution to study drugs. Adverse events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.
Time Frame: Every cycle during treatment (up to 14 cycles)
Population: Since only two participants were accrued, patient confidentiality prevents the reporting of these two participants.
Arm/Group | DC-APCC
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Prostate-cancer Specific Mortality
Time Frame: Registration to Prostate-cancer specific mortality (Up to 3 years)
Population: Since only two participants were accrued, patient confidentiality prevents the reporting of these two participants.
Arm/Group | DC-APCC
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Prostate-specific Antigen (PSA) Progression
Description: In patients whose PSA has not decreased, progressive disease is a 25% increase over the baseline (on-study) and an increase in the absolute-value PSA level by at least 5 ng/mL, which is confirmed by a second value. In patients whose PSA has decreased but has not reached response criteria, progressive disease would be considered to have occurred when PSA increases 25% over the nadir, provided that the increase is a minimum of 5 ng/mL and is confirmed.
  The start of the time to PSA progression is the day treatment is initiated. If at least a 50% decline in PSA has been achieved, the end date is the time the PSA has increased 50% above the nadir at a minimum of 5 ng/mL (this is the same as the parameter for PSA response). For patients without a PSA decrease of this magnitude (or no decrease in PSA), the end point for progression will be calculated at the time a 25% increase in PSA has been achieved (see above). All end dates require a confirmatory PSA.
Time Frame: Registration to PSA progression (Up to 3 years)
Population: Since only two participants were accrued, patient confidentiality prevents the reporting of these two participants.
Arm/Group | DC-APCC
Number analyzed (Participants) | 0

5. Secondary Outcome: Duration of PSA-based Response
Description: PSA-based response was defined as a PSA decline of at least 50%, which must be confirmed by a second PSA value in 4 or more weeks later.
  The duration of PSA-based response are measured from the first time point at which the PSA has declined by at least 50% (which must eventually be confirmed by a second value) until PSA has increased back to 50% of the original on-study value.
Time Frame: Up to 3 years
Population: Since only two participants were accrued, patient confidentiality prevents the reporting of these two participants.
Arm/Group | DC-APCC
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in Quality of Life (QOL) as Measured by the EORTC QLQ-C30 Questionnaire
Description: European Orgnisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-C30 for cancer patients composed of 5 functional scales, 3 symptom scales, a global health status QOL scale, and six single items. Scores for each scale/item were calculated according to the questionnaire's scoring algorithm and range in 0 to 100, with high score represents high healthy level of functioning, high QOL or high level of symptomatology/problems. Change: Scores at cycle 1 minus scores at baseline.
  Change from baseline in QOL will also be evaluated at cycle 6, 10, 15 and every 6 months during observation phase.
Time Frame: Baseline and cycle 1
Population: Since only two participants were accrued, patient confidentiality prevents the reporting of these two participants.
Arm/Group | DC-APCC
Number analyzed (Participants) | 0

7. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS based on radiographic criteria was defined as the time from registration to the time of radiographic progression. A confirmed progression was defined as one for which radiological evidence of a new lesion is found following CT and/or bone scans.
Time Frame: Up to 3 years
Population: Since only two participants were accrued, patient confidentiality prevents the reporting of these two participants.
Arm/Group | DC-APCC
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Since only two participants were accrued, patient confidentiality prevents the reporting of these two participants.
Arm/Group | DC-APCC
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes